CLINICAL TRIAL: NCT02718118
Title: A Prospective, Randomized, Multi-Center, Subject- and Evaluator-Blinded, Parallel Comparison of Dysport®, When Reconstituted at 1.5 mL and 2.5 mL, for the Treatment of Moderate to Severe Glabellar Lines.
Brief Title: Comparison of Dysport Reconstitution at 1.5 mL and 2.5 mL for the Treatment of Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US10348
Record Dates: First submitted 2016-03-16; First posted 2016-03-24 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2018-09

CONDITIONS: Glabellar Lines; Wrinkles
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.5 mL Reconstitution (Experimental): Subjects treated with Dysport reconstituted at 1.5 mL (0.05 mL/injection) following the US on-label guidelines, with each subject receiving a single treatment session (50 units [U]) at the Day 1 visit.
  Interventions: Device: Dysport reconstituted at 1.5 mL (0.05 mL/injection)
- 2.5 mL Reconstitution (Experimental): Subjects treated with Dysport reconstituted at 2.5 mL (0.08 mL/injection) following the US on-label guidelines, with each subject receiving a single treatment session (50 units [U]) at the Day 1 visit.
  Interventions: Device: Dysport reconstituted at 2.5 mL (0.08 mL/injection)

INTERVENTIONS:
Device: Dysport reconstituted at 1.5 mL (0.05 mL/injection) — Subjects treated for moderate to severe (GLSS = 2 or 3) glabellar lines at maximum frown.
  Arms: 1.5 mL Reconstitution
Device: Dysport reconstituted at 2.5 mL (0.08 mL/injection) — Subjects treated for moderate to severe (GLSS = 2 or 3) glabellar lines at maximum frown.
  Arms: 2.5 mL Reconstitution

SUMMARY:
This study is designed to evaluate the safety, efficacy, and subject and investigator satisfaction of 2 different injection volumes of Dysport in the glabellar lines.

1. To determine the proportion of composite responders (based on blinded evaluator and subject assessments) who achieve at least a 1-point reduction from baseline in glabellar line severity score (GLSS) at maximum frown line on Day 30.
2. To assess the GLSS, at maximum frown and at rest, by live assessment at all visits.
3. To evaluate the onset of effect on appearance of glabellar lines starting at the Day 2 visit (subject and blinded evaluator).
4. To assess the subject's satisfaction with the treatment.
5. To evaluate investigator satisfaction of treatment outcome.
6. To evaluate subject psychological well-being.
7. To evaluate subject age appraisal.
8. To evaluate all adverse events during the course of the study.

DETAILED DESCRIPTION:
Five month, randomized, subject- and evaluator-blinded, multi-center, mult-visit study. Subjects treated with Dysport following the US on-label guidelines.

ELIGIBILITY:
Key Inclusion Criteria:

1. Botulinum toxin naïve subject (facial area)
2. Moderate to severe (GLSS = 2 or 3) glabellar lines at maximum frown and mild to severe (GLSS = 1, 2, or 3) glabellar lines at rest using the validated 4-point Photographic Scale, as assessed by the treating investigator and the blinded evaluator.

Key Exclusion Criteria:

1. Have known allergies or sensitivities to Dysport®, any of its excipients, or cow's milk protein
2. Have rhytids of the glabellar region that cannot be smoothed out by manually spreading the skin apart
3. Have a history or have signs and symptoms of eyelid or brow ptosis or signs of compensatory frontalis muscle activity, as judged by the investigator
4. Have clinical or subclinical neuromuscular junctional disorders (eg, myasthenia gravis, Lambert Eaton syndrome, or amyotrophic lateral sclerosis) or a history of dysphagia or aspiration
5. Are women who are pregnant or breast-feeding or who intend to get pregnant within the duration of the study
6. Have an active inflammation or infection in the areas to be treated or had any prior surgery, tattoos, piercings, or scarring in the facial area that, in the opinion of the investigator, may interfere with the results
7. Have had any previous insertion of any permanent or semi-permanent material, hyaluronic acid, or collagen fillers in the glabellar region
8. Have any chronic or acute medical condition that, may pose a risk to the safety of the subject, or may interfere with the assessment of safety or efficacy in this study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Mashburn, PhD, Study Director — Galderma Laboratories, LP
Locations (3):
- United States (3):
  - AboutSkin Dermatology and DermSurgery, Greenwood Village, Colorado
  - Skin Research Institute, Coral Gables, Florida
  - Marina Peredo, MD, PC, Smithtown, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Started | 30 | 30
Completed | 28 | 29
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (10.93) | 46.5 (11.73) | 45.8 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 29 | 29 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Composite Responders Who Achieve at Least a 1-point Reduction From Baseline in Glabellar Line Severity Score (GLSS) at Maximum Frown.
Description: Proportion of composite responders who achieve at least a 1-point reduction from baseline in glabellar line severity score (GLSS) based on subject and blinded-evaluator assessment of glabellar line severity at maximum frown on Day 30.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 27 | 26

2. Secondary Outcome: Proportion of Responders, at Maximum Frown (Subject)
Description: Proportion of responders, at maximum frown, with GLSS at least 1-point reduction from baseline on days 2, 3, 4, 7, 14, 30, 90 and 120 based on assessments by subject using a static 4-point categorical (subject) scale.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 14 | 17

3. Secondary Outcome: Proportion of Responders, at Maximum Frown (Blinded Evaluator)
Description: Proportion of responders, at maximum frown, with GLSS at least 1-point reduction from baseline on days 2, 3, 4, 7, 14, 30, 90 and 120 based on assessments by blinded evaluator using a validated 4-point photographic scale.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 21 | 20

4. Secondary Outcome: Proportion of Responders, at Maximum Frown (Treating Investigator)
Description: Proportion of responders, at maximum frown, with GLSS at least 1-point reduction from baseline on days 2, 3, 4, 7, 14, 30, 90 and 120 based on assessments by treating investigator using a validated 4-point photographic scale.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 19 | 16

5. Secondary Outcome: Proportion of Combination Responders, at Maximum Frown (Blinded Evaluator and Subject)
Description: Proportion of combination responders, at maximum frown, with GLSS at least 1-point reduction from baseline on days 2, 3, 4, 7, 14, 30, 90 and 120 based on assessments made by blinded evaluator and subject.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 13 | 14

6. Secondary Outcome: Proportion of Responders, at Rest (Subject)
Description: Proportion of responders, at rest, with GLSS at least 1-point reduction from baseline on days 2, 3, 4, 7, 14, 30, 90 and 120 based on assessments made by subject using a static 4-point categorical (subject) scale.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 20 | 18

7. Secondary Outcome: Proportion of Responders, at Rest (Blinded Evaluator)
Description: Proportion of responders, at rest, with GLSS at least 1-point reduction from baseline on days 2, 3, 4, 7, 14, 30, 90 and 120 based on assessments made by blinded evaluator using a validated 4-point photographic scale.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 14 | 14

8. Secondary Outcome: Proportion of Responders, at Rest (Treating Investigator)
Description: Proportion of combination responders, at rest, with GLSS at least 1-point reduction from baseline on days 2, 3, 4, 7, 14, 30, 90 and 120 based on assessments made by treating investigator using a validated 4-point photographic scale.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 17 | 17

9. Secondary Outcome: Proportion of Combination Responders, at Rest (Blinded Evaluator and Subject)
Description: Proportion of combination responders, at rest, with GLSS at least 1-point reduction from baseline on days 2, 3, 4, 7, 14, 30, 90 and 120 based on assessments made by blinded evaluator and subject.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 9 | 10

10. Secondary Outcome: Proportion of Subjects Who Achieved an Onset of Effect on the Appearance of the Subject's Glabellar Lines.
Description: Combination endpoint from both subject and blinded evaluator assessments. Assessments made on days 2, 3, 4, and 7.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 28 | 28

11. Secondary Outcome: Subject Satisfaction With the Treatment of Glabellar Lines - I am Satisfied With How I Look.
Description: Proportion of subjects who responded 'agree' or 'strongly agree' regarding change from baseline in subject satisfaction questionnaire on day 120.
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 19 | 20

12. Secondary Outcome: Investigator Satisfaction With Treatment Outcome - Satisfied With the Study Product Results
Description: Proportion of treating investigators who responded 'agree' or 'strongly agree' to the individual satisfaction questions on Day 30.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
Participants | 29 | 26

13. Secondary Outcome: Subject Psychological Well-being - Mean Change at Day 120 Compared to Baseline
Description: Mean change from baseline on day 120 using the Psychological Well-Being (FACE-Q).Total score for entire questionnaire is transformed to a Rasch score, scale of 0-100.
  Increase in score = increased well-being.
Time Frame: Baseline and Day 120
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
score on a scale | 28.6 (32.93) | 20.3 (31.02)

14. Secondary Outcome: Subject Age Appraisal Using the FACE-Q-Age Appraisal Visual Analog Scale (VAS) - Mean Change at Day 120 Compared to Baseline
Description: Mean change from baseline on day 120 using the FACE-Q Age Appraisal VAS. "0" years represents "current age subjects rated their appearance as older or younger than current age"; "+" years represents "older than current age"; "-" years represents "younger than current age".
Time Frame: Baseline and Day 120
Measure: Mean (Standard Deviation); unit: years
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
years | -3.0 (7.59) | -4.6 (5.94)

15. Secondary Outcome: Subject Appraisal of Lines Between the Eyebrows (FACE-Q) - Mean Change at Day 120 Compared to Baseline
Description: Mean change from baseline on day 120 using the Subject Appraisal Lines Between the Eyebrows (FACE-Q).Total score for entire questionnaire is transformed to a Rasch score, scale of 0-100. Increase in score = less bothered by glabellar lines.
Time Frame: Baseline and Day 120
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
Number analyzed (Participants) | 30 | 30
score on a scale | 33.9 (33.14) | 30.4 (24.70)

ADVERSE EVENTS:
Time Frame: 120 days
Arm/Group | 1.5 mL Reconstitution | 2.5 mL Reconstitution
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.5 mL Reconstitution (N=30) | 2.5 mL Reconstitution (N=30)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No